CLINICAL TRIAL: NCT00144508
Title: An Open-Label, Phase III Study to Evaluate the Efficacy and Safety of MRA in Patients With RA
Brief Title: Phase III Comparative Study(Open-Label) of MRA for Rheumatoid Arthritis(RA)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chugai Pharmaceutical (Industry)
Responsible Party: Chugai Pharmaceutical, Chugai Pharmaceutical
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MRA012JP
Record Dates: First submitted 2005-09-02; First posted 2005-09-05 (Estimated); Last update posted 2009-02-02 (Estimated); Status verified 2009-01

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: MRA (Tocilizumab)
- 2 (Other): continue current treatment
  Interventions: Other: current treatment

INTERVENTIONS:
Drug: MRA (Tocilizumab) — 8mg /kg /4week for 52 weeks
  Arms: 1
Other: current treatment — continue current treatment
  Arms: 2

SUMMARY:
To evaluate clinical efficacy and tolerability of MRA, patients with RA are randomized to receive either MRA or conventional DMARDs.

ELIGIBILITY:
Inclusion criteria

* Diagnosed as having RA, on the basis of the criteria stipulated by the American Conference on Rheumatism (ACR) in 1987.
* With RA that has continued for at least 6 months but less than 5 years, with the date of first appearance being taken as the date of RA diagnosis.
* Active RA despite at least one DMARD or immunosuppressant. Active disease is defined as having at least 6 tender and 6 swollen joints among 49 and 46 joints stipulated by the Japanese Rheumatism Foundation's Drug Evaluation Committee and ESR at least 30 mm/hr and CRP not less than 2.0mg/dL.

Exclusion criteria

* Shown to have class-IV Steinbrocker's functional activity in an evaluation carried out within 4 weeks before administration of the study drug.
* Treated with drugs that delay joint destruction (infliximab, etanercept, leflunomide, etc.) within 3 months before administration of the study drug.
* The oral corticosteroid dose (prednisolone equivalent of up to 10 mg/day)has not been fixed 2 weeks before administration of the study drug.
* Subjected to any of the following within 4 weeks before administration of the study drug: (i) Change in dosage of currently administered DMARDs and/or immunosuppressive agents. (ii) Plasma exchange method. (iii) Surgical treatment (operations, etc.).

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Actual)
Dates: Start 2003-03; Primary Completion 2004-05 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Change in the erosion score, as determined by the modified Sharp method. | week 52
Frequency and severity of adverse events and adverse drug reactions | throughout study

SECONDARY OUTCOMES:
Change in the erosion score | week 28
Changes in the joint space narrowing score and total Sharp score | week 28, 52

CONTACTS AND LOCATIONS:
Overall Officials: Takahiro Kakehi, Study Director — Chugai Pharmaceutical